CLINICAL TRIAL: NCT06379022
Title: Clinical and Cellular Responses of Tissues at Newly Restored Single Implants Compared to Contralateral Natural Teeth During Their First Year of Functional Loading
Brief Title: Proteomic Analysis of Newly Restored Single Implants
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Danae A. Apatzidou, Associate Professor, Aristotle University Of Thessaloniki
Other Study IDs: AUTh-29/21-11-2018
Record Dates: First submitted 2024-04-18; First posted 2024-04-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Peri-Implantitis; Peri-implant Mucositis; Periodontal Diseases
Keywords: Peri-implant tissue; tissue remodeling; first year of function; proteomics; crevicular fluid; periodontal parametres
MeSH Terms: conditions — Peri-Implantitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Samples of crevicular fluid collected from the periodontal and the peri-implant crevice
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Implant unit: Newly restored single implant that is closely followed for plaque control
  Interventions: Behavioral: Plaque control
- Tooth unit: A contralateral tooth that is closely followed for plaque control
  Interventions: Behavioral: Plaque control

INTERVENTIONS:
Behavioral: Plaque control — Subjects are motivated for optimal oral hygiene

SUMMARY:
In 10 systemically healthy non-smokers, free of periodontitis, one newly restored implant (baseline-T0) and one corresponding tooth were followed over 12 months (T1). All implants were screw-retained, and platform-switched. Oral hygiene was closely monitored during the study. Probing pocket depth (PPD), attachment levels (CAL), bleeding and plaque indices and crevicular fluid were collected from an implant-site (PICF) and a tooth-site (GCF). Total proteomic profiles in PICF and GCF were investigated using label-free quantitative proteomics.

DETAILED DESCRIPTION:
Study population A total of 10 systemically healthy non-smokers, who were previously treated for periodontal disease and received implant therapy, were recruited between December 2018 and November 2019. Each subject contributed with a newly restored screw-retained implant 2-4 weeks following functional loading (baseline, T0) and was closely followed over 12 months (T1). All study implants were platform-switched (ø4.1. Straumann® Bone Level) and were installed following a two-stage surgical placement protocol. A contralateral tooth in the same jaw, but on the opposite quadrant, served as the control. Implant placement was planned based on clinical and cone beam computerized tomography evaluations and was performed using a prosthetic guide. Implants were submerged and were exposed 6 months later when a healing abutment was adjusted on the fixture followed by a screw-retained crown 1 month later. Exclusion criteria included younger than 18 years of age, <18 teeth (excluding third molars), untreated periodontal disease, periodontitis Stage III-IV, evidence of peri-implantitis (Berglundh et al, 2018) at other implant sites, significant soft tissue pathology, untreated carious cavities (five or more), systemic diseases that require intake of medications, medical conditions that contraindicated surgical implant placement, the medication that interferes with bone metabolism, pregnancy or lactation, inadequate dimensions of the alveolar ridge or grafted bone at the surgical site, and tooth extraction 3 months prior to the study, smoking.

Clinical assessments Site-specific and full-mouth clinical indices were assessed at T0 and T1. Oral hygiene instructions using a manual toothbrush and the modified Bass technique were re-iterated at four time points over the 12-month study period (T0, 3-, 6-months and T1). Prophylaxis comprising supragingival ultrasonic debridement and polishing with a rubber cup was carried out at the same time points. In detail, the following site-specific clinical indices probing pocket depth (PPD), clinical attachment levels (CAL), recession (REC), modified gingival index (MGI) (score range 0-4) (Lobene et al. 1986), modified dental plaque index (mPI)1 (score range: 0-3) and modified sulcus bleeding index (mBI)1 (score range: 0-3) were determined at the mesial buccal site of the study implant in a similar manner as PPD, CAL, REC, MGI, plaque index (PI)2 (score range: 0-3) and sulcus bleeding index (SBI)3 (score range: 0-5) at the control tooth site. The width of keratinized tissues (KTW) was determined at the mid-buccal aspect of the test-implant/control tooth. Moreover, on a full-mouth basis PPD, CAL and dichotomous supragingival dental plaque (PI) (O'Leary et al., 1972) and bleeding on probing (BOP) (Ainamo et al., 1975) were recorded at six sites per tooth/implant present in the mouth. Periodontal clinical indices were determined using a manual periodontal probe (PCP-UNC 15; Hu-Friedy XP-23/QW, Hu-Friedy, Chicago, IL, USA) to the nearest millimeter.

Radiographic examination The VixWin™ Platinum Gendex software (Hatfield, PA, USA) linearly assessed the distance between the implant platform and the bone crest (I-BC) parallel to the long axis of the implant fixture at T0 and T1 on intra-oral digital radiographs. Periapical digital radiographs (RadioVisioGraphy; Trophy Radiology S.A., Paris, France) were obtained using the long cone paralleling technique at a 10 cm distance between the x-ray head and the digital sensor.

Collection of crevicular fluid samples Peri-implant crevicular fluid (PICF) was collected from the mesial-buccal site of the newly restored study implant, while gingival crevicular fluid (GCF) was collected from the mesial-buccal site of a contralateral control tooth at T0 and T1. Before PICF/GCF collection, the surfaces were gently air-dried and isolated from saliva by placing cotton rolls and using a saliva ejector. Then, supragingival plaque was carefully removed by sterile curettes and paper strips (Periopaper, OraFlow Inc., Smithtown, NY, USA) were gently placed in the mesial aspect of the peri-implant/gingival sulcus until mild resistance was felt and held for 30 sec. Care was taken to avoid mechanical trauma when placing the strips and those strips contaminated with blood were discarded. The strips were stored in Eppendorf tubes (Eppendorf, Hamburg, Germany) at -80C until further processed.

Proteomic analysis of crevicular fluid samples (PICF/GCF) The PICF and GCF samples collected from the study implant sites (n=10) and the control tooth sites (n=10), respectively at T0 and T1 were pooled and used for proteomics analysis. In brief, 20 µg of total protein per pooled sample were reduced, alkylated, trypsinized, and purified with single-pot, solid-phase-enhanced sample preparation (SP3) assisted protein digestion using the PreOmics' SP3-iST (PreOmics GmbH) following the manufacturing protocol for protein extraction and digestion. These extracts were concentrated using a Speedvac (Thermo Savant SPD121P, Thermo Scientific, Waltham, MA, USA) and stored at -20 °C until further use.

The digested samples were first reconstituted with 30 µL of 3% acetonitrile (ACN) in 0.1% formic acid then subjected to Fusion Orbitrap Lumos mass spectrometer (Thermo Fisher Scientific) interfaced to an Easy nano-flow HPLC system (Thermo Fisher Scientific) for proteomics analysis. During proteomics analysis, a three-liner gradient of acetonitrile and water was used with 0.1% formic acid at a 300 nL/minute flow rate. The gradient progressed from 2% to 30% acetonitrile over 60 minutes, then from 30% to 97% acetonitrile in 10 minutes, and finally held at 97% acetonitrile for 10 minutes. The mass spectrometer was set to operate in a data-dependent manner, automatically switching between MS and MS/MS using the Xcalibur software package from Thermo Fisher Scientific. A mass range of 300-1500 m/z was selected for the Orbitrap analyzer.

The acquired MS data were processed using the Mascot (version 2.4.1, Matrix Science) search engine against an in-house database containing 10,125,458 entries, which included human (accessed on 22nd February 2022 from Uniprot) and bacterial (accessed on 22nd February 2022 from eHOMD) proteins, common MS contaminants, and reverse sequences for estimating the false discovery rate. During the proteomics analysis, the precursor ion tolerance and fragment ion tolerance were set to 10 ppm and ±0.6 Da, respectively. Up to two missed cleavages per peptide were allowed for tryptic digestion. The carbamidomethylation modification on cysteine was selected as a fixed modification, while deamidation of asparagine and glutamine and oxidation of methionine were chosen as variable modification parameters.

The spectrum reports of the search results were generated using Scaffold software (version 4.2.1, Proteome software), and proteins with FDR at 1%, minimal 2 unique peptides identified, as peptide FDR at 0.1% were used for relative protein abundance analysis. Fold changes in abundance intensity were calculated based on value log2 fold change (FC) between pairs of consecutive time points using R-software (R: A Language and Environment for Statistical Computing, R Development Core Team). Proteins with a log2FC ≥ 1 of unique spectrum counts between two conditions or exclusively identified in one condition were considered regulated.

Bioinformatics analysis for the regulated proteins The regulated proteins underwent overrepresentation analysis (ORA) against the Hallmark database using the WebGestalt online tool. The analysis, conducted on March 25th, 2022, aimed to compare the regulation of proteins in teeth and implants between T0 and T1 conditions. Similarly, on March 29th, 2022, the analysis examined the regulation of proteins in both teeth and implants under either the T0 or T1 conditions. The top 10 enriched results, ranked by p-value using the hypergeometric distribution, were reported. However, only pathways with a p-value < 0.05 were considered as regulated.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy non-smokers having a single implant prosthetically restored (2-4 weeks).

Exclusion Criteria:

* younger than 18 years of age, <18 teeth (excluding third molars), untreated periodontal disease, periodontitis Stage III-IV, evidence of peri-implantitis (Berglundh et al, 2018) at other implant sites, significant soft tissue pathology, untreated carious cavities (five or more), systemic diseases that require intake of medications, medical conditions that contraindicated surgical implant placement, the medication that interferes with bone metabolism, pregnancy or lactation, inadequate dimensions of the alveolar ridge or grafted bone at the surgical site, and tooth extraction 3 months prior to the study, smoking.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — self reported if not overt
Study Population: Systemically healthy non-smokers, who were previously treated for periodontal disease and recently received implant therapy; Each subject contributed with one newly restored screw-retained implant 2-4 weeks following functional loading (baseline, T0) and was closely followed over 12 months (T1).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-11-29 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth | baseline and 12 months
  Assessed by a periodontal probe
Protein expression | baseline and 12 months
  proteomic analysis

SECONDARY OUTCOMES:
Recession | baseline and 12 months
  Assessed by a periodontal probe
Bleeding upon probing | baseline and 12 months
  Assessed after probing teh crevice
Inflammation index | baseline and 12 months
  Assessed visually

CONTACTS AND LOCATIONS:
Overall Officials: Danae A Apatzidou, Assoc. Professor, Study Chair — Dental School, Aristotle University; Danae A Apatzidou, Assoc. Professor, Principal Investigator — Dental School, Aristotle University
Locations (1):
- Dental School, Aristotle University, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No
Available upon request

REFERENCES:
- [Derived] Apatzidou DA, Violesti A, Konstantinidis A, Bao K, Silbereisen A, Bostanci N. Protein profile at newly restored implants compared to contralateral teeth over 12-months: a pilot study. Clin Oral Investig. 2024 Oct 11;28(11):590. doi: 10.1007/s00784-024-05984-w. PMID 39390228